CLINICAL TRIAL: NCT03368534
Title: Autologous Regenerative Technology (ART) For Wound Healing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Device needs modifications
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Geoffrey C. Gurtner, Professor of Surgery, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 42628
Record Dates: First submitted 2017-11-27; First posted 2017-12-11 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Chronic Wounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Skin Wound Patients (Experimental): Patients will receive ART for wound healing and will be followed for 28 days to determine success of the procedure.
  Interventions: Device: Autologous Regenerative Technology (ART)

INTERVENTIONS:
Device: Autologous Regenerative Technology (ART) — ART device with single-needle, fluid-assisted skin tissue harvesting technology.

SUMMARY:
The purpose of the study is to provide a more effective method of harvesting skin with minimal or no pain, heal more rapidly with little scarring in an outpatient setting with the use of only local anesthesia.

DETAILED DESCRIPTION:
Skin wounds sometimes are difficult to heal by primary closure and often require tissue substitution by autologous grafting requiring harvesting of donor skin. The latter may cause morbidities such as risk of infection, discoloration, pain, and scarring of both donor and recipient areas. Full-thickness stin grafts (FTSG) are created when the entire dermis and epidermis are harvested, These grafts are typically used for acute full-thickness wounds where the wound can sustain and nourish the graft and improved cosmesis is important. Split-thickness skin grafting (STSG) has been used to close large skin wounds, and it involves the harvesting of the epidermis and upper dermis from a donor site. It is generally the preferred grafting method for restoring the structural integrity of chronic wounds, as the wound bed may not have the ability to support a FTSG. Nevertheless, because deep dermal structures such as sweat glands and hair follicles are not harvested, the STSG is functionally abnormal. Before the grafting process takes place, STSGs are commonly meshed and enlarged, increasing the coverage area and allowing fluid drainage. However, the meshing process produces a "fish-net" appearance of the grafted skin. Other limitations include healing of the donor site, which often is delayed and leaves unappealing pigmentary changes and, at times, scar formation.

Currently, engineered "off the shelf" grafts such as cadaveric skin, xenografts, and artificial skin substitutes are being used in the management of chronic, difficult to heal wounds. Skin substitutes work by providing cells, growth factors, and other key elements that promote healing while preventing extracellular matrix degradation. However, these only offer transient wound coverage, and require secondary healing of the wound itself. Thus, autologous skin grafting continues to be necessary. Scar formation at the donor and grafted site remain most troublesome morbidities in autologous skin grafting. Scar tissue is stiff, dysfunctional, often painful, and tends to contract over time, producing skin irregularities.

In contrast, skin remodeling is a process that substitutes missing tissue while preserving tissue architecture. While scarring is triggered by large-scale tissue damage, remodeling is stimulated by microscopic tissue damage. This principle became clear when fractional photothermolysis (FP) was developed that is currently used for photoaged skin treatment and wound scars. In FP, laser microbeams are used to produce microscopic thermal injury per cm2 of skin surface, which causes very thin columns of tissue damage or ablation. It has been found that columns less than 500 µm in diameter heal promptly without scarring. FP involves full-thickness (i.e. complete epidermis and dermis) tissue injury in which the epidermis closes within 1 day, and the dermal damage is fixed in around 2 weeks, followed by tissue remodeling without scarring.

Because the experience with FP showed that millions of small, full-thickness columns of skin tissue can be removed without scarring, it was hypothesized that full-thickness microscopic skin tissue columns (MSTCs) could be harvested from healthy skin with insignificant donor site-morbidity and that these MSTCs could function as a graft to accelerate wound healing.

To explore this, a prototype device was developed that can harvest hundreds of full-thickness columns of skin tissue (500 micrometer diameter) using single-needle, fluid-assisted harvesting technology. The harvested MSTCs can subsequently be placed directly onto a wound to aid in healing.

With conventional full thickness grafts and split thickness grafts, the donor area requires sometimes a period of immobility, requiring attentive wound care and pain management. The ART may provide a more effective method of harvesting skin with minimal or no pain, healing rapidly with little scarring. This can take place in an outpatient setting, with the use of only local anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Any age ranging 18-90, any gender or ethnic background is a candidate.
* Subjects with chronic wounds that have been present for at least 4 weeks

Exclusion Criteria:

* Pregnant women.
* Adults unable to consent.
* Prisoners.
* Subjects requiring concurrent systemic antimicrobials during the study period for any infection.
* Subjects with leg lesions and clinically significant and unreconstructed peripheral arterial disease.
* Subjects who are receiving immunosuppressive agents, radiation therapy, or cytotoxic agents.
* Subjects who require treatment for a primary or metastatic malignancy (other than squamous or basal cell carcinoma of the skin).
* Subjects with other conditions considered by the investigator to be reasons for disqualification that may jeopardize subject safety or interfere with the objectives of the trial (e.g., acute illness or exacerbation of chronic illness, lack of motivation, history of poor compliance).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Patient-reported pain at skin donor site at Day 7 | Day 7
  Pain will be assessed on an 11-point visual analogue scale (range 0 to 10, with 0 corresponding to no pain, and 10 corresponding to the worst pain imaginable)
Patient-reported pain at skin donor site at Day 14 | Day 14
  Pain will be assessed on an 11-point visual analogue scale (range 0 to 10, with 0 corresponding to no pain, and 10 corresponding to the worst pain imaginable)
Patient-reported pain at skin donor site at Day 21 | Day 21
  Pain will be assessed on an 11-point visual analogue scale (range 0 to 10, with 0 corresponding to no pain, and 10 corresponding to the worst pain imaginable)
Patient-reported pain at skin donor site at Day 28 | Day 28
  Pain will be assessed on an 11-point visual analogue scale (range 0 to 10, with 0 corresponding to no pain, and 10 corresponding to the worst pain imaginable)
Patient-reported tolerability of ART procedure | End of study (Day 28)
  Tolerability will be assessed on an 10-point scale (range 1 to 10, with 1 corresponding to most tolerable, and 10 corresponding to least tolerable)
Physician-reported tolerability of ART procedure | End of study (Day 28)
  Tolerability will be assessed on an 10-point scale (range 1 to 10, with 1 corresponding to most tolerable, and 10 corresponding to least tolerable)
Percent change in size of wound area as a measure of time to healing at Day 7 | Day 7
Percent change in size of wound area as a measure of time to healing at Day 14 | Day 14
Percent change in size of wound area as a measure of time to healing at Day 21 | Day 21
Percent change in size of wound area as a measure of time to healing at Day 28 | Day 28
Time to full epithelialization as a measure of quality of healing | Baseline to Day 28
  Epithelialization is defined as growth of epithelium over the wound surface

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey Gurtner, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Advanced Wound Care Center, Redwood City, California, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share data